CLINICAL TRIAL: NCT00521443
Title: Cryosurvival of Embryos From Dysmorphic Oocytes
Status: Completed | Type: Observational
Sponsor: V.K.V. American Hospital, Istanbul (Other)
Other Study IDs: AH-05/04
Record Dates: First submitted 2007-08-24; First posted 2007-08-27 (Estimated); Last update posted 2007-08-27 (Estimated); Status verified 2007-08

CONDITIONS: Cryopreservation; Blastocyst
MeSH Terms: interventions — Cryopreservation

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

GROUPS / COHORTS (12):
- Normal: Embryos derived from morphologically normal MII oocytes
  Interventions: Procedure: Cryopreservation, thawing and blastocyst culture
- Irregular Shapes: Embryos derived from irregularly shaped oocytes.
  Interventions: Procedure: Cryopreservation, thawing and blastocyst culture
- Large PVS: Embryos derived from oocytes with large perivitelline space.
  Interventions: Procedure: Cryopreservation, thawing and blastocyst culture
- Dark Zona: Embryos derived from oocytes with dark zona pellucida
  Interventions: Procedure: Cryopreservation, thawing and blastocyst culture
- Dark cytoplasm: Embryos derived from oocytes with dark cytoplasm
  Interventions: Procedure: Cryopreservation, thawing and blastocyst culture
- Vacuolar cytoplasm: Embryos derived from oocytes with vacuolated cytoplasm
  Interventions: Procedure: Cryopreservation, thawing and blastocyst culture
- Central granulation: Embryos derived from oocytes with centrally granulated cytoplasm
  Interventions: Procedure: Cryopreservation, thawing and blastocyst culture
- Double extra: Embryos derived from oocytes with double extracytoplasmic abnormalities
  Interventions: Procedure: Cryopreservation, thawing and blastocyst culture
- Double combined: Embryos derived from oocytes with any combination of one extracytoplasmic and one cytoplasmic anomaly
  Interventions: Procedure: Cryopreservation, thawing and blastocyst culture
- Double cytoplasmic: Embryos derived from oocytes with any two cytoplasmic anomalies
  Interventions: Procedure: Cryopreservation, thawing and blastocyst culture
- Triple extra: Embryos derived from oocytes with triple extracytoplasmic anomaly
  Interventions: Procedure: Cryopreservation, thawing and blastocyst culture
- Triple combined: Embryos derived from oocytes with triple combined anomalies
  Interventions: Procedure: Cryopreservation, thawing and blastocyst culture

INTERVENTIONS:
Procedure: Cryopreservation, thawing and blastocyst culture — Good quality human embryos were frozen - thawed and cultured to the blastocyst stage.

SUMMARY:
Various morphological abnormalities of human oocytes were reported to detrimentally affect embryo development. We observed development of frozen thawed embryos derived from oocytes with normal or abnormal morphological features to the blastocyst stage. Cytoplasmic abnormalities of the oocytes were found to negatively affect cryosurvival potential of the embryos.

ELIGIBILITY:
Inclusion Criteria:

* Human embryos derived from morphologically normal or abnormal mature oocytes that fertilized normally by microinjection procedure.
* Embryos were obtained from couples who refused to freeze their supernumerary embryos after fresh embryo transfer in an assisted reproduction treatment cycle.

Exclusion Criteria:

* Embryos obtained after microinjection to immature oocytes taht were in vitro matured in culture.
* Embryos obtained from abnormally fertilized zygotes.

Ages: 18 Years to 45 Years | Sex: Female
Age Groups: Adult

CONTACTS AND LOCATIONS:
Overall Officials: Basak Balaban, B.Sc., Study Director — Assisted Reproduction Unit of the VKV American Hospital of Istanbul
Locations (1):
- VKV American Hospital, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Derived] Balaban B, Ata B, Isiklar A, Yakin K, Urman B. Severe cytoplasmic abnormalities of the oocyte decrease cryosurvival and subsequent embryonic development of cryopreserved embryos. Hum Reprod. 2008 Aug;23(8):1778-85. doi: 10.1093/humrep/den127. Epub 2008 May 12. PMID 18477573